CLINICAL TRIAL: NCT00823797
Title: A Phase II Study of Bendamustine in the Treatment of Recurrent High-Grade Gliomas (Anaplastic Gliomas and Glioblastoma)
Brief Title: Bendamustine Hydrochloride in Treating Patients With Recurrent or Progressive Anaplastic Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Maciej Mrugala, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6803; NCI-2010-00714 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 6803 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bendamustine hydrochloride) (Experimental): Patients receive bendamustine hydrochloride IV over 30-90 minutes on days 1-2. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bendamustine Hydrochloride; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Bendamustin Hydrochloride; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treanda
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well bendamustine hydrochloride works in treating patients with anaplastic glioma or glioblastoma that has come back (recurrent) or growing, spreading or getting worse (progressive). Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary endpoint for this study is the 6-month progression-free survival-i.e., the proportion of patients who remain alive and free of any tumor progression at 6 months.

SECONDARY OBJECTIVES:

I. To determine the safety of single agent bendamustine (Treanda) (bendamustine hydrochloride) the treatment of malignant gliomas.

II. To determine the efficacy of bendamustine (Treanda) as a single agent as assessed by progression-free survival (PFS) at 6 months.

III. To assess quality of life using the Functional Assessment of Cancer Therapy-Brain (FACT-BR).

OUTLINE:

Patients receive bendamustine hydrochloride intravenously (IV) over 30-90 minutes on days 1-2. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 2 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have had prior pathologic confirmation of tumor histology, anaplastic glioma (AG) or glioblastoma (GBM) and have supratentorial gliomas
* Patients must have shown unequivocal evidence for tumor recurrence or progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan with contrast
* The recurrence to be treated needs to be the 1st or 2nd recurrence of the AG or GBM
* If a patient has had surgery prior to enrolling on study, an enhanced MRI or CT scan should be done within 96 hours prior to surgery or at least 4-6 weeks after surgery
* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

  * They are > 2 weeks from surgery
  * They have recovered from the effects of surgery
  * Evaluable or measurable disease following resection of recurrent tumor is mandated for eligibility into the study
  * To best assess the extent of residual disease post-operatively, an enhanced CT/MRI should be done no later than 96 hours after surgery or it will need to be done 4-6 weeks post-operatively; if the 96 hour scan is more than 2 weeks from registration, the scan needs to be repeated
* A baseline scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for at least 5 days otherwise a new baseline MR/CT is required; the same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement
* Patients must have failed prior external beam radiation therapy; a positron emission tomography (PET) or thallium single photon emission computed tomography (SPECT), MR spectroscopy and MR perfusion, or surgical documentation may be done at the discretion of the treating physician if there is a question of radiation changes/necrosis versus progressive disease
* Stereotactic radiosurgery (SRS):

  * Patients must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium SPECT, MR spectroscopy and MR perfusion or surgical documentation of disease
  * At least 12 weeks between completion of SRS and initiation of bendamustine
* Interstitial brachytherapy: patients must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium SPECT, MR spectroscopy and MR perfusion or surgical documentation of disease
* Patients must have had at least one prior chemotherapy regimen that included temozolomide and no more than one prior salvage chemotherapy
* Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least 2 weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count), 4 weeks for experimental biologic agents (epidermal growth factor receptor [EGFR] inhibitors, etc) and 7 weeks from Gliadel implantation
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must sign an authorization for the release of their protected health information
* Patients must have a life expectancy > 11 weeks
* Patients must have a Karnofsky performance status of > 60
* White blood cells (WBC) >= 3,000/ul
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 80,000/mm^3
* Hemoglobin >= 9 mg/dl (NOTE: eligibility level for hemoglobin may be reached by transfusion)
* Absolute lymphocyte count >= 200/mm^3
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) < 3 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Serum creatinine < 1.5 mg/dL
* Calculated creatinine, glomerular filtration rate (GFR) >= 30 cc/minute

Exclusion Criteria:

* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Known human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible
* Patients must not be pregnant or breast feeding and must practice adequate contraception
* Patients can only be on non-enzyme inducing anti-convulsants; if they are on an enzyme inducing anti-convulsant, they may be converted to a non-enzyme inducing anticonvulsants
* Patients cannot be taking any cytochrome P450, cytochrome P450, family 1, subfamily A, polypeptide 2 (CYP1A2) pathway inhibiting or inducing agents (except proton pump inhibitors which are allowed) including cimetidine, antidepressants, antibiotics and all others
* Known sensitivity to bendamustine
* Known sensitivity to mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2015-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Mrugala, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma: Anaplastic Glioma Arm
  Patients receive bendamustine hydrochloride IV over 30-90 minutes on days 1-2. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
- Treatment (Bendamustine Hydrochloride) for Glioblastoma: Glioblastoma Arm
  Patients receive bendamustine hydrochloride IV over 30-90 minutes on days 1-2. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma | Treatment (Bendamustine Hydrochloride) for Glioblastoma
Started | 29 | 16
Completed | 29 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma | Treatment (Bendamustine Hydrochloride) for Glioblastoma | Total
Number analyzed (Participants) | 29 | 16 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 13 | 41
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 17 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 16 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 26 | 14 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: PFS-6
Description: Defined as the proportion of patients who remain alive and free of any disease progression at 6 months. PFS over time will be estimated using the Kaplan-Meier method with standard errors estimated using Greenwood's formula.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bendamustine Hydrochloride) for Glioblastoma | Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma
Number analyzed (Participants) | 16 | 29
Participants | 1 | 8

2. Secondary Outcome: PFS
Description: Defined as the time from date of initial therapy to first objective documentation of tumor progression or death.
Time Frame: Up to progression or death, whichever came first, assessed up to 108 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bendamustine Hydrochloride) for Glioblastoma | Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma
Number analyzed (Participants) | 16 | 29
months | 1.0 [-0.5 to 2.6] | 2.6 [-1.0 to 6.3]

3. Secondary Outcome: Toxic Death
Description: Defined as death that is possibly, probably, or definitely attributed to bendamustine hydrochloride.
Time Frame: Up to 30 days after completion of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bendamustine Hydrochloride) for Glioblastoma | Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma
Number analyzed (Participants) | 16 | 29
Participants | 0 | 0

4. Secondary Outcome: Overall Survival
Description: *inclusive of subjects still alive at time of last reporting.
Time Frame: Until death or last reported survival
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Bendamustine Hydrochloride) for Glioblastoma | Treatment (Bendamustine Hydrochloride) for Anaplastic Glioma
Number analyzed (Participants) | 16 | 29
months | 18.3 [8.2 to 28.4] | 45.6 [33.6 to 57.7]

ADVERSE EVENTS:
Arm/Group | Treatment (Bendamustine Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 3/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bendamustine Hydrochloride) (N=45)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic Reaction (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bendamustine Hydrochloride) (N=45)
Lymphopenia (Blood and lymphatic system disorders) | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No